CLINICAL TRIAL: NCT07256990
Title: Development of Adaptive Intervention for Early Detection and Management of Chronic Kidney Disease in Syria
Brief Title: An e-Learning Program for Nurses on Evidence-Based Prevention of CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Fatema Ahmed, Principal Investigator, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-R-091
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Nursing Education
Keywords: e-learning; nurses; CKD prevention; Syria; pilot study; pre-post; professional development

STUDY DESIGN:
Intervention Model Description: Single-arm pilot; all eligible nurses receive the same e-learning programme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-learning group (Experimental): All eligible nurses receive the 7-module asynchronous e-learning programme on evidence-based CKD prevention.
  Interventions: Behavioral: CKD-prevention e-learning course (Your Kidney... our priority)

INTERVENTIONS:
Behavioral: CKD-prevention e-learning course (Your Kidney... our priority) — 'Seven online modules (videos, infographics, case studies, quizzes) delivered via Google Classroom over 4 weeks. Content covers CKD risk-factor screening, lifestyle & dietary counselling, co-morbidity management, patient education, and program evaluation. Each module includes a short lecture (<12 min), interactive case, downloadable poster, and 5-item quiz (pass ≥75 %). Participants can download materials for offline use.'

SUMMARY:
Electronic training course to help Syrian nurses prevent chronic kidney disease Why are the investigators doing this study? Chronic kidney disease (CKD) is common in Syria, yet many nurses have not received up-to-date training on early detection or patient education for risk reduction. The investigators aim to determine whether a brief, phone-friendly online course can improve nurses' knowledge, day-to-day practice, confidence, and satisfaction.

What will happen? Registered nurses employed in nephrology, cardiology, or endocrinology units will be invited to participate.

Each nurse will complete a short online quiz and questionnaire before the course.

Participants will then work through seven brief learning modules (videos, posters, case stories, quizzes) on a phone or computer over four weeks.

Two weeks after the final module, participants will repeat the same quiz and questionnaire so the investigators can measure any change.

The investigators will also request feedback on course acceptability and suggestions for improvement.

Possible benefits If the course proves effective, the investigators plan to offer it to additional nurses across Syria and distribute the materials free of charge.

Number of volunteers the investigators plan to enrol 30 nurses (single group; no randomisation). Primary outcome the investigators will measure Change in CKD-prevention knowledge score from baseline to immediately post-course.

DETAILED DESCRIPTION:
Study design Prospective, single-arm, pre-test/post-test pilot trial to estimate preliminary effect, feasibility, and acceptability of a seven-module asynchronous e-learning programme on Syrian hospital nurses' CKD-prevention knowledge, self-reported practice, confidence, and satisfaction. No control or randomization will be used.

Setting & recruitment Thirty registered nurses employed in nephrology, cardiology, or endocrinology wards of Syrian hospitals will be recruited through convenience sampling (hospital WhatsApp groups, professional associations, social-media promotion). Inclusion criteria: (1) registered nurse license, (2) access to smartphone/tablet, (3) willingness to provide electronic informed consent. A dedicated WhatsApp group will be created for announcements and technical support only; no teaching will occur in this group.

Intervention development Content was constructed by the study team and refined through a two-round Delphi panel (two nephrologists, two nutritionists, one senior nurse). Modules map to 2022 KDIGO prevention guidelines and WHO self-care recommendations. All assets (slide-casts ≤ 12 min, branching case vignettes, infographic posters, patient hand-outs) will be bilingual (Arabic/English subtitles) and compressed to ≤ 25 MB to allow offline download.

Delivery logistics Google Classroom will release two modules per week for four weeks. Each module contains: (1) voiced micro-lecture or animation, (2) interactive case study with branched questions, (3) downloadable poster & patient hand-out, (4) 5-item quiz (pass mark 75 %; unlimited attempts). Engagement analytics (views, quiz attempts, offline downloads) will be extracted from the Google Workspace admin console. Participants will receive a 5 USD mobile-data stipend to mitigate connectivity barriers; no other incentive will be offered.

Data collection timeline Day 0 - Baseline Qualtrics link (demographics, 38-item CKD-knowledge scale, 7-item attitude, 5-item practice, 24-item confidence).

Weeks 1-4 - Intervention delivered. Week 6 - Post-intervention Qualtrics link (same instruments plus 30-item E-Learning Satisfaction Questionnaire and one open-ended feedback item).

No biological samples or patient-level data will be collected. Outcomes Primary: change in CKD-prevention knowledge score (0-38; KR-20 = 0.83). Secondary: change in attitude (7-item, 5-point Likert, CVI = 0.89), self-reported practice (5-item, test-retest r = 0.78), confidence (24-item, Cronbach α = 0.92); module-quiz performance (% correct, attempts to pass); overall satisfaction (0-100; α = 0.93 Arabic version); qualitative feedback (inductive thematic analysis, two independent coders, κ target > 0.80).

Sample size Thirty participants will be enrolled. This number meets pilot-guidance (≥ 30) to detect a large within-group effect (Cohen's d ≥ 0.8) and allows 15 % attrition.

Analysis plan Normality will be examined with Shapiro-Wilk tests. Pre-post differences will be analysed using Wilcoxon signed-rank tests (two-tailed, α = 0.05). Effect size will be reported as r (Z/√N) and Cohen's d with 95 % CIs. Feasibility benchmarks: recruitment ≥ 80 % of target within four weeks, module-completion ≥ 70 %, mean satisfaction ≥ 4/5. Qualitative data will follow Braun & Clarke six-step thematic analysis.

Ethics & dissemination Approvals obtained from Shandong University IRB (No. 2023-R-091) and Tishreen University IRB (Ref. N14218). Electronic informed consent will be secured; withdrawal permitted at any time without penalty. Data will be stored on password-protected Qualtrics and OneDrive (256-bit AES). Findings will be submitted to a peer-reviewed journal and presented at nephrology/nursing-education conferences. De-identified dataset and e-learning package will be shared on reasonable request after publication.

ELIGIBILITY:
Inclusion Criteria:

1. Registered nurse currently employed in a Syrian hospital
2. Works in nephrology, endocrinology, or cardiology ward
3. Age 18 - 60 years
4. Has smartphone or computer access with internet connection
5. Willing to complete pre- and post-course questionnaires
6. Provides electronic informed consent

Exclusion Criteria:

1. Not a registered nurse (e.g., nursing assistant, student)
2. Outside the specified age range
3. Unable to access online materials (no device / no internet)
4. Previous participation in the same e-learning pilot
5. Refuses to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-21 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Change in CKD-prevention knowledge score from baseline to immediately post-intervention | Baseline and Week 6
  38-item multiple-choice quiz; score range 0-38; higher score indicates better knowledge.

SECONDARY OUTCOMES:
Change in self-reported practice | Baseline and Week 6
  5-item Likert scale (1-5); total score 5-25.
Change in confidence level | Baseline and Week 6
  24-item Likert scale (1-5); total score 24-120.
Change in attitude toward CKD prevention | Baseline and Week 6
  7-item Likert scale (1-5); total score 7-35.
Overall satisfaction with the e-learning programme | Week 6
  30-item validated satisfaction scale (0-100 %).
Module quiz performance | After each of the 7 modules (Weeks 1-4)
  Percentage of correct answers per 5-item quiz.

CONTACTS AND LOCATIONS:
Overall Officials: Kefang Wang, PhD, Study Director — Shandong University , School of Nursing and Rehabilitation
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data for knowledge, practice, confidence, attitude, and satisfaction scores, together with the study protocol and analytic code, will be made available to researchers who provide a methodologically sound proposal approved by the corresponding author. Data will be shared via a secure, password-protected cloud link for 5 years after publication. Proposals should be directed to fatema92w@gmail.com
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months after the publication of primary results and ending 5 years post-publication
Access Criteria: Researchers must submit a scientifically relevant proposal, sign a data-use agreement, and use the data only for non-commercial research. Ethical approval may be required